CLINICAL TRIAL: NCT04342949
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Study to Investigate the Auxiliary Effects of Fucoidan in Patients With Locally Advanced Rectal Cancer Who Receive Combined Radio-chemotherapy Before Surgery
Brief Title: The Auxiliary Effects of Fucoidan for Locally Advanced Rectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Vice Superintendent, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUHIRB-F(I)-20180113
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: To Observe Whether the Fucoidan Can Improve the Quality of Life of the Such Patients Receiving the Neoadjuvant CCRT
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: quality of life — To observe the difference of quality of life

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel study. The main goal is to investigate the auxiliary effects of Fucoidan for the patients with locally advanced rectal cancer who receive neoadjuvant CCRT before surgery. The quality of life is our primary endpoint for this study. The study is an observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Age was more/equal to 20 year-old and less/equal to 80 year-old
2. Diagnosed as locally advanced rectal cancers by pathological biopsy and image study.
3. ECOG performance status within 0 to 2 points
4. Excepted life remaining at least 4 months
5. Females with fertility are willing to use effective contraception during the period of study
6. Willing to follow the test procedures and tracking procedures
7. sign the inform consent form

Exclusion Criteria:

1.Suffering from other primary malignant tumors 2.Females who are pregnant, planning to become pregnant, or breastfeeding 3.Participate in other interventional clinical trial within the first 30 days 4.Suffering from major mental illness such as mental retardation and mental disorders 5.Unable to understand and answer research questions (oral or written) 6.Abnormal laboratory data within 14 days before joining the study 7.Evidence that subject has a severe or uncontrolled disease

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we enrolled the patients with locally advanced rectal cancers and received neoadjuvant CCRT (concurrent radiochemotherapy) before.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
auxiliary effects of Fucoidan | 2 years
  To evaluate the quality of life after unblind by 4th edit of FACT-C

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, Ph.D, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsai HL, Yeh YS, Chen PJ, Chang YT, Chen YC, Su WC, Chang TK, Huang CW, Wang JY. The Auxiliary Effects of Low-Molecular-Weight Fucoidan in Locally Advanced Rectal Cancer Patients Receiving Neoadjuvant Concurrent Chemoradiotherapy Before Surgery: A Double-Blind, Randomized, Placebo-Controlled Study. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231187153. doi: 10.1177/15347354231187153. PMID 37822243